CLINICAL TRIAL: NCT05789641
Title: Role of Dynamic Contrast-enhanced Ultrasound (D-CEUS) and 2D Elastography in the Evaluation of Portal Hypertension and Risk of Oesophageal Variceal Bleeding in Patients With Liver Cirrhosis
Brief Title: Multimodal Ultrasound and Portal Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Zocco Maria Assunta, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2986
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to international guidelines, Hepatic Venous Pressure Gradient is the gold standard technique for portal hypertension measurement, but it is invasive and poorly available. Currently, surveillance of oesophageal/gastric varices is performed by upper gastrointestinal endoscopy. More recently, non-invasive tools to estimate portal hypertension have been developed and, among them, ultrasound elastography has been proposed as a technique to stratify patient risk to have portal hypertension.

Aim of this study is to evaluate the relationship between ultrasound evaluation (D-CEUS + elastography) and endoscopic parameters predictive of clinically significant portal hypertension in patients with liver cirrhosis.

DETAILED DESCRIPTION:
Background: About 80-90% of cirrhotic patients shows portal hypertension signs, including ascites, splenomegaly, oesophageal and/or gastric varices, encephalopathy. According to international guidelines, Hepatic Venous Pressure Gradient is the gold standard technique for portal hypertension measurement, but it is invasive and poorly available. Currently, surveillance of oesophageal/gastric varices is performed by upper gastrointestinal endoscopy. More recently, non-invasive tools to estimate portal hypertension have been developed and, among them, ultrasound elastography has been proposed as a technique to stratify patient risk to have portal hypertension. More specifically, liver stiffness <20kPa together with platelet count > 150.000/m3 (Baveno VI criteria) or > 100.000/mm3 (Expanded Baveno VI criteria) are considered at low risk of portal hypertension. D-CEUS provides information about microvascularization and it is widely used to characterize focal liver lesions, but recent data show its role also in evaluating the degree of liver fibrosis and portal hypertension.

Primary objective: To evaluate the relationship between ultrasound evaluation (D-CEUS + elastography) and endoscopic parameters predictive of clinically significant portal hypertension in patients with liver cirrhosis.

Secondary objectives:

* To identify quantitative ultrasound parameters able to predict the presence of clinically significant portal hypertension.
* To identify cut-off values of ultrasound parameters able to stratify the risk of bleeding in patients with oesophageal varices
* To evaluate the relationship between the hemodynamic changes induced by endoscopic and/or pharmacological therapy of oesophageal varices highlighted with ultrasound (D-CEUS + elastography) and the hemodynamic changes highlighted by endoscopy.

Study design: Single-centre prospective observational study Methods: consecutive adult patients with liver cirrhosis needing to undergo endoscopic evaluation of portal hypertension will be enrolled in the Unit of Internal Medicine and Gastroenterology of the Policlinico Agostino Gemelli. Cirrhotic patients of different aetiologies will be included. Exclusion criteria will be previous recent endoscopic treatment of oesophageal varices (<6 months), portal and/or splanchnic thrombosis, portal cavernomatosis, acute or chronic heart failure, previous liver transplantation, presence of hepatocellular carcinoma or other hepatic neoplasms, inadequate visualization of the liver parenchyma on B-mode ultrasound, known allergy to ultrasound contrast medium, pregnancy and lactation. Assuming a disagreement rate of 5% between ultrasonographic and endoscopic diagnosis and considering an α=0.05 and a power of 90%, a sample size of N=73 patients is calculated. Patients will undergo ultrasound (B-mode, shear-wave elatography and D-CEUS) and endoscopic evaluation (diagnostic esophagogastroduodenoscopy plus endoscopic treatment of eosophageal or gastric varices, if needed) as per clinical practice. After obtaining informed consent, personal, clinical and laboratory data will be collected and analysed specifically for the study.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age more than 18 years
* diagnosis of cirrhosis of different etiologies

Exclusion criteria:

* previous recent endoscopic treatment of oesophageal varices (<6 months)
* portal and/or splanchnic thrombosis
* portal cavernomatosis
* acute or chronic heart failure
* previous liver transplantation
* presence of hepatocellular carcinoma or other hepatic neoplasms
* inadequate visualization of the liver parenchyma on B-mode ultrasound
* known allergy to ultrasound contrast medium
* pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult cirrhotic patients
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
to evaluate the relationship between ultrasound and endoscopic parameters which predict clinically significant portal hypertension | 3 months after endoscopic exam

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy